CLINICAL TRIAL: NCT01894594
Title: Alkali Therapy in Subjects With Sickle Cell Disease (SCD) - Evaluation of Efficacy, Safety, and Beneficial Effects
Brief Title: Efficacy, Safety Study and Benefit of Alkali Therapy in Sickle Cell Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Jane Little, Director, Sickle Cell Disease Program, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-12-13
Record Dates: First submitted 2013-07-03; First posted 2013-07-10 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2018-02

CONDITIONS: Sickle Cell Anemia; Chronic Kidney Disease; Metabolic Acidosis
Keywords: Sickle cell disease; Chronic kidney disease; Bicarbonate therapy
MeSH Terms: conditions — Anemia, Sickle Cell; Renal Insufficiency, Chronic; Acidosis | interventions — Sodium Bicarbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sodium Bicarbonate (Experimental): Patients will be monitored at baseline bi-weekly intervals for 12 weeks, the first 4 weeks to establish a stable baseline, followed by 8 weeks of alkali therapy, as follows:
  Interventions: Drug: Sodium Bicarbonate

INTERVENTIONS:
Drug: Sodium Bicarbonate — Oral sodium bicarbonate tablets administered at a starting dose of 0.6 mEQ/Kg body weight and will be escalated once, at 4 weeks, to 0.9 mEQ/Kg body weight.
  Weekly schedule:
  0-4 weeks: Serial Measurement at baseline, without therapy 4-8 weeks: *~0.6 mEq/kg of ideal body weight of Sodium Bicarbonate tablets divided into TID dosing 8-12 weeks: *~0.9 mEq/kg of ideal body weight of Sodium Bicarbonate tablets divided into TID dosing
  * to the closest dose of 650 mg (7.74 mEq)
  Ideal Body Weight is defined by the following formulas (Devine Calculation):
  Ideal Body Weight (men) = 50 + 2.3 (Height (in) - 60) Ideal Body Weight (women) = 45.5 + 2.3 ( Height (in) - 60)
  Other Names: Alkali Therapy

SUMMARY:
The objective of this study is to assess the effect of alkali administration on bicarbonate and potassium levels in patients with Sickle Cell Disease (SCD) and depressed serum bicarbonate levels. The study is a prospective non-blinded evaluation of tolerability and efficacy of alkali repletion with 4 weeks of observation and two sequential 4 week courses of escalating oral sodium bicarbonate treatment.

DETAILED DESCRIPTION:
Primary Objective:

To assess the effect of alkali administration on bicarbonate and potassium levels in patients with SCD and depressed serum bicarbonate levels.

Secondary Objectives:

To assess the effect of alkali administration on improvement in hemolysis and on sequelae of impaired kidney function, ie, LDH, Hgb, reticulocyte count, red cell half-life, and muscle strength, Vitamin D levels, and markers of bone turnover, respectively.

To assess the influence of alkali administrations on markers of kidney tubule inflammation.

To evaluate intraparenchymal iron in patients with SCD and renal dysfunction. Safety and adverse events of alkali patients with sickle cell disease will be monitored. This research will supplement current knowledge about management of the clinically important subset of people with SCD who have renal insufficiency and acid-base perturbation.

ELIGIBILITY:
Inclusion Criteria:

* Sickle cell disease patients with HbSS
* eGFR <90 ml/min/1.73m2 (determined by abbreviated 4 variable modification MDRD equation) and/or measured urinary albumin to creatinine ratio >30mg/g.
* Age ≥18 years

Exclusion Criteria:

* Previous chronic treatment with alkali (including sodium bicarbonate, calcium carbonate or baking soda)
* Bicarbonate level >25 mEq/L
* Decompensated heart failure
* Uncontrolled systolic blood pressure >140 mm/Hg (the cutoff for systolic hypertension in SCD is lower than in non-SCD)
* Moderate-to-severe lower extremity edema
* Projected progression to ESRD within 6 months
* Kidney transplantation
* Treatment with immunosuppressives within the last 3 months
* Vasoocclusive (VOC) within 1 week of study entry
* Active (open) leg ulcer
* Change in hydroxyurea dose within the last 3 months, unless a self-limited interruption of a stable dose
* Blood transfusion within 8 weeks, unless on chronic transfusions
* Pregnancy
* Inability to give informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-06; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Serum bicarbonate level | 12 weeks
  To assess the effect of alkali administration on bicarbonate and potassium levels in patients with SCD and depressed serum bicarbonate levels.

SECONDARY OUTCOMES:
Hemolysis markers | 12 weeks
  To assess the effect of alkali administration on improvement in hemolysis and on sequelae of impaired kidney function, ie, LDH, Hgb, reticulocyte count, red cell half-life, and muscle strength, Vitamin D levels, and markers of bone turnover, respectively.

OTHER OUTCOMES:
Tubular effect | 12 weeks
  To assess the influence of alkali administrations on markers of kidney tubule inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Jane Little, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University hospitals Case Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No